CLINICAL TRIAL: NCT00661752
Title: Quarter-Time Myocardial Perfusion SPECT
Brief Title: Protocol for Evaluation of Quarter-Time Cardiac Imaging: 5-Minutes Rest and 3-Minutes Stress Wide Beam Reconstruction (WBR) Versus Full-Time Filtered Back Projection (FBP)
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: E.Gordon DePuey, MD, St.Luke's-Roosevelt Hospital Center
Other Study IDs: quarter-time cardiac SPECT
Record Dates: First submitted 2008-04-08; First posted 2008-04-18 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Cardiac Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- FBP studies: standard filtered backprojection image processing/reconstruction of full-time acquisition data
  Interventions: Device: quarter-time stress scans reconstructed by WBR (4SPS) - Xpress3.Cardiac; Device: quarter-time rest scans reconstructed by WBR (6/8/10 SPS) - Xpress3.Cardiac
- half-time WBR: wide-beam reconstruction of simulated half-time acquisitions from standard full-time acquisitions
  Interventions: Device: quarter-time stress scans reconstructed by WBR (4SPS) - Xpress3.Cardiac; Device: quarter-time rest scans reconstructed by WBR (6/8/10 SPS) - Xpress3.Cardiac
- Quarter-time stress: 4 seconds per stop post-stress SPECT acquisitions reconstructed by the wide-beam reconstruction method
  Interventions: Device: quarter-time stress scans reconstructed by WBR (4SPS) - Xpress3.Cardiac
- Quarter-time rest: 6 seconds per stop rest SPECT acquisitions reconstructed by the wide-beam reconstruction method
  Interventions: Device: quarter-time rest scans reconstructed by WBR (6/8/10 SPS) - Xpress3.Cardiac

INTERVENTIONS:
Device: quarter-time stress scans reconstructed by WBR (4SPS) - Xpress3.Cardiac — Comparison of the diagnostic quality of quarter-time WBR stress with stress studies generated via FBP and half-time WBR
  Other Names: WBR; wide-beam reconstruction; Xpress3.Cardiac
  Groups: FBP studies; Quarter-time stress; half-time WBR
Device: quarter-time rest scans reconstructed by WBR (6/8/10 SPS) - Xpress3.Cardiac — Comparison of the diagnostic quality of 6 SPS quarter-time rest acquisitions with FBP and half-time WBR rest studies; simulated 8 SPS and 10 SPS quarter-time rest acquisitions are also compared to FBP and half-time WBR rest studies.
  Other Names: WBR; wide-beam reconstruction; Xpress3.Cardiac
  Groups: FBP studies; Quarter-time rest; half-time WBR

SUMMARY:
A new, innovative software image processing method, wide beam reconstruction (WBR), utilizes resolution recovery and incorporates Poisson noise-reduction into the reconstruction process of NM images. This method facilitates the reconstruction of low count density myocardial perfusion SPECT images. Preliminary research indicates that SPECT acquisition time consequently can be reduced by 60% (less than 5 minutes) for rest and by 75% (just over 3 minutes) for stress, while tomographic image quality is maintained, or even improved. Such a decrease in image acquisition time decreases patient discomfort during the tomographic acquisition, decreases the opportunity for patient motion, and improves laboratory efficiency.

DETAILED DESCRIPTION:
Standard full-time SPECT will be processed using FBP and compared to 3-minute stress and 5-minute rest scans processed with WBR. The following scan parameters will be evaluated: image quality; perfusion defect extent, severity, and reversibility; transient ischemic dilatation; left ventricular end-diastolic volume; left ventricular end-systolic volume; left ventricular ejection fraction; and regional wall motion and wall thickening abnormalities. These parameters will be assessed visually by experienced Nuclear physicians (at least 2 blinded readers) and quantitatively using several different commercially available software programs.

ELIGIBILITY:
Inclusion Criteria:

* Patient is clinically stable
* Patient is able to tolerate additional 8 minutes of scanning
* Patient is willing to undergo additional 8 minutes of scanning

Exclusion Criteria:

* Unstable patient
* Non-consenting patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients referred to St. Luke's NM lab. for clinically indicated myocardial perfusion SPECT
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Image quality of quarter-time WBR images is equivalent/superior to full-time FBP | March 2008

SECONDARY OUTCOMES:
Image quality of quarter-time WBR is equivalent/superior to half-time WBR | March 2008

CONTACTS AND LOCATIONS:
Overall Officials: Gordon DePuey, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center